CLINICAL TRIAL: NCT04565847
Title: The Effects of Salbutamol on Mannitol Induced Cough Responses in Healthy Controls
Acronym: COMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Gail Gauvreau, Professor Department of MEdicine, McMaster University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: McMaster-COMA-11537
Record Dates: First submitted 2020-08-17; First posted 2020-09-25 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Cough
MeSH Terms: conditions — Cough | interventions — Albuterol; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: albutamol or placebo will be delivered following a mannitol cough challenge in a randomized, double-blind crossover design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Control - Active Arm (Active Comparator): Healthy Controls Mannitol-Induced Cough Challenges on Visit 2 to determine elligibility (cough response). Mannitol delivered via inhalation. Dosage: 0, 5, 10, 20, 40 mg capsules. 80 and 160 mg doses delivered with two and four capsules, respectively. Nebulized salbutamol (5mg/mL) given prior to Mannitol-Induced Cough Challenges on Visit 3 or 4.
  Interventions: Drug: Salbutamol 5mg/mL
- Healthy control - Placebo Arm (Placebo Comparator): Healthy Controls Mannitol-Induced Cough Challenges on Visit 2 to determine elligibility (cough response). Mannitol delivered via inhalation. Dosage: 0, 5, 10, 20, 40 mg capsules. 80 and 160 mg doses delivered with two and four capsules, respectively. Nebulized 0.9% Saline given prior to Mannitol-Induced Cough Challenges on Visit 3 or 4.
  Interventions: Drug: Sodium Chloride 0.9% Inhl 3Ml

INTERVENTIONS:
Drug: Salbutamol 5mg/mL — Nebulized salbutamol given prior to Mannitol-Induced Cough Challenge
  Other Names: Ventolin nebuliser
  Arms: Healthy Control - Active Arm
Drug: Sodium Chloride 0.9% Inhl 3Ml — Nebulized 0.9% saline given prior to Mannitol-Induced Cough Challenge
  Other Names: Placebo Comparator
  Arms: Healthy control - Placebo Arm

SUMMARY:
The study aim is to investigate if changes in osmolarity using mannitol challenge can evoke coughing healthy controls with no evidence of bronchoconstriction (PC20>16mg/ml or mannitol PD15 > 635 mg, or < 10% incremental fall in FEV1 between consecutive mannitol doses) and if salbutamol can affect this. This is a double-blind, placebo-controlled analysis in healthy controls assessing the effects of salbutamol on mannitol induced cough.

DETAILED DESCRIPTION:
The study will have a maximum of 4 visits separated by at least 24 hours. The first 2 visits will determine eligibility. All eligible subjects will be invited back for a third and a fourth visit.

Screening Period (Visits 1 and 2) - For All Subjects Eligible subjects will be identified during the initial screening procedures with measures of spirometry, hyperresponsiveness to methacholine, complete history, physical examination, allergen skin test, and mannitol cough challenge. The screening procedures will be conducted over 2 separate visits.

Effects of Salbutamol (Visit 3 and 4) - For Healthy Control Subjects, Twenty subjects with no evidence of asthma will return for visit 3 and 4. These visits must be at least 24h apart and no longer than 7 days. Health controls will first receive salbutamol 2.5mg or saline placebo via a nebuliser and 15 mins later the forced expiratory volume at one second (FEV1) measured. Subjects will then undergo a mannitol cough challenge exactly like the previous mannitol cough challenges. These data will be used for determining the effects of salbutamol on mannitol-induced cough.

Visit Windows Each visit must be separated by a minimum of 24 hours, and a maximum of 7 days. Study visits can be performed in the morning or afternoon, however for each subject the timing should be consistent with Visits 2 at the same time of day ± 2 hours

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and give written informed consent.
2. Male and female volunteers 18 through 65 years of age.
3. No airway hyperresponsiveness as determined by methacholine PC20>16mg/ml or mannitol PD15 > 635 mg, or < 10% incremental fall in FEV1 between consecutive mannitol doses.
4. Fall in FEV1 of ≤ 5% after any mannitol dose during mannitol challenge compared to baseline FEV1 at 0 mg at screening mannitol challenge (Visit 2).
5. Baseline FEV1≥ 80% of the predicted value.
6. Demonstrate cough response to inhaled mannitol.

Exclusion Criteria:

1. Current or former smoker with >10-pack-year history
2. Current or previous history of other significant respiratory disease
3. Significant systemic disease, including history of current malignancy or autoimmune disease
4. Pregnancy or breastfeeding.
5. Use of corticosteroids within 28 days prior to the first study visit.
6. Use of nonsteroidal anti-inflammatory drugs (NSAIDs) within 48 hours of study visits or aspirin with 7 days of study visits
7. Use of antihistamines including those in cold and allergy medications within 72 hours of study visits
8. Use of caffeine-containing products within 4 hours of study visits
9. Use of ACE inhibitors
10. Any centrally acting medication which in the view of the investigator could alter the sensitivity of the cough reflex including but not restricted to tricyclic anti-depressants, pregabalin, gabapentin, codeine, tramadol, or any other opioid.
11. Unwillingness or inability to comply with the study protocol for any other reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Primary Outcome - Emax | Through study completion, an average of 1 year
  The effect of salbutamol on mannitol induced coughs Emax - the maximum number of coughs at any dose of mannitol.

SECONDARY OUTCOMES:
Cough dose response curves | Through study completion, an average of 1 year
  Comparison of mannitol-induced cough dose response curves in normal healthy controls treated with salbutamol compared with placebo.
ED50 | Through study completion, an average of 1 year
  The effect of salbutamol on mannitol induced coughs E50 - the dose of mannitol causing half the maximal response.
C2 | Through study completion, an average of 1 year
  Comparison of the mannitol dose causing 2 coughs (C2) in a mannitol induced cough challenge in healthy controls treated with salbutamol compared with placebo.
C5 | Through study completion, an average of 1 year
  Comparison of the mannitol dose causing 5 coughs (C5) in a mannitol induced cough challenge in healthy controls treated with salbutamol compared with placebo.
Cumulative number of coughs | Through study completion, an average of 1 year
  Comparison of the cumulative number of coughs in a mannitol induced cough challenge in healthy controls treated with salbutamol compared with placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Gail Gauvreau, PhD, Principal Investigator — McMaster University Hospital
Locations (2):
- Canada (2):
  - McMaster Cardio-Respiratory Research Lab, Hamilton, Ontario
  - McMaster University, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No